CLINICAL TRIAL: NCT05158634
Title: Investigation of the Relationship of Trunk Control and Endurance with Balance and Functional Mobility in Children with Cerebral Palsy
Brief Title: Relationship of Trunk Control and Endurance with Balance and Functional Mobility in Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Asena Yekdaneh, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: A.Gulnergiz
Record Dates: First submitted 2021-11-21; First posted 2021-12-15 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2023-12

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Trunk Control; Mobility; Balance; Functional Health; Endurance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cerebral Palsy: Inclusion Criterias: Being diagnosed with Cerebral Palsy. Volunteer. Be between the ages of 6-18. Being at level 1 and level 2 according to Gross Motor Function Classification System (GMFCS) (Level 1 and 2).
  To have the cognitive skills to understand and apply the evaluation parameters.
  Exclusion Criterias: Cognitive impairment of participants diagnosed with Cerebral Palsy. Participants diagnosed with Cerebral Palsy have vision or hearing problems. Participants diagnosed with Cerebral Palsy must have a history of trauma such as botox or muscle relaxation operation and/or fracture at least 6 months before participating in the study.
  Interventions: Other: Evaluations

INTERVENTIONS:
Other: Evaluations — Within the scope of the study, the participants will be evaluated for 30 minutes in a single session. The participants' trunk stabilization and endurance, balance, functional mobility, upper extremity endurance, functional health and quality of life will be questioned by questionnaires, scales and tests. Evaluation will begin with a literature-supported demographic data form prepared for the participants.
  Assessments to be made are listed below. Trunk Control Measurement Scale (TCMS) Pediatric Balance Scale (PBS) Time Up and Go test (TUG) Trunk Flexor Test (TFT) The Pediatric Outcomes Data Collection Instrument (PODCI)

SUMMARY:
It is predicted by studies that the motor and cognitive performance disorders seen in children with Cerebral Palsy (CP) may lead to loss of balance, postural control and mobility. At the same time, trunk muscle fatigue seen in children with CP is a critical motor problem and may cause deficits in adjusting the proper connection between the trunk and pelvis stabilizers.These deficits can lead to impairments in balance, postural control and mobility. Considering the relationship between the deficits seen in children with CP and postural control and postural control with the trunk, the idea that there is a need for studies that evaluate the trunk in every way and reveal its relationship with balance, postural control and mobility in order to organize the rehabilitation program effectively in children with CP. Therefore, in the planning of our study, it was aimed to evaluate trunk control and endurance in children with CP and to examine their relationship with balance and functional mobility parameters, as well as to reveal their relationship with functional health and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Being diagnosed with Cerebral Palsy Volunteer Be between the ages of 6-18 Being at level 1 and 2 according to Gross Motor Function Classification System (GMFCS) (Level 1-2).

To have the cognitive skills to understand and apply the evaluation parameters.

Exclusion Criteria:

Participants diagnosed with Cerebral Palsy having cognitive disorders Participants diagnosed with Cerebral Palsy having vision or hearing problems Participants diagnosed with Cerebral Palsy have a history of trauma such as botox or muscle relaxation operation and / or fracture at least 6 months before participating in the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Being diagnosed with Cerebral Palsy. Being at level 1 and 2 according to Gross Motor Function Classification System (GMFCS) (Level 1-2). Be between the ages of 6-18.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Trunk Control Measurement Scale (TCMS) | Baseline
  TCMS consists of static sitting balance, dynamic sitting control (Selective motor control and dynamic reaching) sections. The scale consists of 15 items in total and is divided into five, seven and three items. All items are evaluated bilaterally and scored on a 2, 3 or 4 point rank scale. TCMS total score is between 0-58 and the higher the score, the better the performance. Participants' trunk stabilization will be evaluated with TCMS.
Pediatric Balance Scale (PBS) | Baseline
  The five-level consists of 14 elements such as sitting balance, standing balance, standing up from sitting, moving from standing to sitting, transfers, stepping, reaching, turning and jumping. Each item is scored between 0-4 points. High scores indicate better performance. Participants' balance will be evaluated with PBS.
Time Up and Go (TUG) | Baseline
  The participant sitting on the floor without arm support, hip and knee flexed at 90 degrees and feet on the ground are asked to stand up, walk 3 meters, turn around and sit on the chair. The test is applied 3 times, the time is recorded and the average of 3 trials is taken. Participants' functional mobility will be evaluated with TUG.
Trunk Endurance | Baseline
  In the test performed to evaluate trunk endurance, the starting position is trunk flexed to 60 degrees (supported by a foam wedge), hips and knees flexed to 90 degrees, and feet in a stable position. In the test position, after the wedge is lifted, the participant is asked to try to keep the body in the flexion position at 60 degrees as much as possible and the time is recorded in seconds. The trunk endurance of the participants will be evaluated with the Trunk Flexor Test.

SECONDARY OUTCOMES:
Modified Push-up Test | Baseline
  In the test used to evaluate the endurance of the upper extremities, in the starting position, individuals are asked to lie in a prone position, take their hands at shoulder level, flex their elbows to the side of the trunk, and bring their knees to 90 degrees of flexion. Then, while in this position, they are asked to raise the head, shoulders and trunk for 30 seconds, with the elbows in full extension. The number of repetitions of the movement for 30 seconds is recorded. Participants' upper extremity endurance will be evaluated with the Modified Push-up Test.
Pediatric Outcomes Data Collection Instrument (PODCI) | Baseline
  PODCI has 2 parent forms (child and adolescent) and adolescent forms consisting of the same questions. The test is a Likert-type scale and consists of 5 parts: Upper Extremity Functions-UEF, Physical Function and Sport-FFS, Transfer and Basic Mobility-TM, Pain-RA and Happiness / Satisfaction-MM, as well as Expectations-TB section where expectations from treatment are questioned. Each section is calculated between 0-100. Participants' quality of life will be evaluated with PODCI.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Asena Yekdaneh, Pt.,MSc., Principal Investigator — Istanbul University - Cerrahpasa
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Universitesi-Cerrahpasa, Istanbul, Istanbul
  - Işıl Özel Eğitim ve Rehabilitasyon Merkezi, Istanbul, Istanbul

IPD SHARING:
Plan to Share IPD: No